CLINICAL TRIAL: NCT07017634
Title: Efficacy and Safety of Novosis Putty in Transforaminal Lumbar Interbody Fusion for Patients With Lumbar Degenerative Disc Disease : A Pivotal, Randomized, Prospective, Multi-Center Study
Brief Title: Efficacy and Safety of NOVOSIS Putty for Interbody Lumbar Fusion Cases
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CGBio Inc. (Industry)
Collaborators: CGBio USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGNVP002
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Novosis Putty (Experimental)
  Interventions: Device: Novosis Putty
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Novosis Putty — Single Level TLIF surgery with Novosis Putty
  Arms: Novosis Putty
Other: Standard of Care — Single Level TLIF surgery with standard of care bone graft
  Arms: Standard of Care

SUMMARY:
Efficacy and Safety of Novosis Putty in Transforaminal Lumbar Interbody Fusion for Patients with Lumbar Degenerative Disc Disease : A Pivotal, Randomized, Prospective, Multi-Center Study

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of symptomatic lumbar degeneration with or without foraminal or recess stenosis of the lumbar confirmed by subject history and radiographic imaging (CT, MRI, X-rays) with no more than a Grade 2 (≤50% translation) spondylolisthesis. Symptomatic lumbar degeneration (L1 to S1) that may be associated with a co-morbid condition.
* Has preoperative Oswestry Disability Index score ≥ 40/100 at baseline
* Psychosocially, mentally and physically able to fully comply with this protocol including adhering to follow-up schedule and requirements and filling out forms
* Signed informed consent

Exclusion Criteria:

* Previous instrumented surgery (i.e.: anterior disc replacement, spinal fusion, interspinous device, etc.) at the index lumbar level or an adjacent level;
* Degenerative or lytic spondylolisthesis greater than Grade 2 (50% translation);
* Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years;
* Any degenerative muscular or neurological condition that would interfere with evaluation of outcomes, including but not limited to Parkinson's disease, amyotrophic lateral sclerosis (ALS), or multiple sclerosis;
* Has chronic or acute renal and/or hepatic impairment and/or failure or prior history of renal and/or hepatic parenchymal disease;
* Lactating, pregnant or interested in becoming pregnant in the next 3 years;
* Is currently participating in an investigational therapy (device and/or pharmaceutical) within 30 days prior to entering the study or such treatment is planned during the 24 months following enrollment into the study.
* Known hypersensitivity or allergy to any components of the study treatments inclusive of hypersensitivity or allergy to any BMP-2 type recombinant proteins or peptides.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Success | 24 months after surgery
  Meet all of the following conditions:
  1. Fusion success
  2. Oswestry Disability Index success
  3. Neurological success
  4. No subsequent surgical interventions
  5. No related serious event

SECONDARY OUTCOMES:
Overall Success | 6 and 12 months after surgery
  Meet all of the following conditions:
  1. Fusion success
  2. Oswestry Disability Index success
  3. Neurological success
  4. No subsequent surgical interventions
  5. No related serious event
ODI score | 6weeks, 3, 6, 12, 24, 36, 48 and 60months after surgery
  Evaluate Oswestry Disability Index(ODI) score/ lowest 0(best) to highest 100(worst)
VAS score | 6weeks, 3, 6, 12, 24, 36, 48 and 60months after surgery
  Evaluate Visual Analog Scale(VAS) score/ none (0 mm) to an extreme amount of pain (100mm)
SF-12 score | 6weeks, 3, 6, 12, 24, 36, 48 and 60months after surgery
  Evaluate SF-12 scores / lowest 0(worst) to highest 100(best)
Intraoperative variables | Intraoperative
  Surgery time, blood loss